CLINICAL TRIAL: NCT06080828
Title: Transdermal Neuromodulation for Management of Chronic Pelvic Pain in Women: A Randomized Placebo-controlled Trial
Brief Title: Transdermal Neuromodulation for Management of Chronic Pelvic Pain in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Kadry, Associate Professor of Physical Therapy, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T/WH/2/2023/42e
Record Dates: First submitted 2023-10-08; First posted 2023-10-12 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Pelvic Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (SG) (Experimental): they will receive treatment with 20 minutes of neuromodulation of the posterior tibial nerve of both lower limbs using Physio Go-lite electrical stimulation device (made by ASTAR, ver 1.0.2 in Poland). Using TENS current in the device, the positive electrode will be placed posterior to the medial ankle malleolus, and the negative electrode will placed ten centimeters away on the leg along the tibial nerve path. The TENS current parameters will be 200 micro second pulse width, 10 Hz frequency, and intensity according to participant tolerance ranging between (10 - 50 mA) that increased gradually until visible movement in the big toe or fanning of toes will be noticed. The therapy sessions will be given three times a week, every other day, for a total of twelve sessions. Alos, they will receive leaflet with information for home instructions on how to properly walk, sleep, maintain good posture, and deal with activities of daily living.
  Interventions: Device: Percutaneous Posterior Tibial Nerve Stimulation; Behavioral: Home instructions
- control group (CG) (Placebo Comparator): They will receive placebo neuromodulation of the posterior tibial nerve in both lower limbs, much as those in the research group. Alos, they will receive leaflet with information for home instructions on how to properly walk, sleep, maintain good posture, and deal with activities of daily living.
  Interventions: Device: Placebo Percutaneous Posterior Tibial Nerve Stimulation; Behavioral: Home instructions

INTERVENTIONS:
Device: Percutaneous Posterior Tibial Nerve Stimulation — 20 minutes of neuromodulation of the posterior tibial nerve of both lower limbs using Physio Go-lite electrical stimulation device (made by ASTAR in Poland, ver 1.0.2 in Poland). Using Transcutaneous Electrical Nerve Stimulation (TENS) current in the device, the positive electrode will be placed posterior to the medial ankle malleolus, and the negative electrode will placed ten centimeters away on the leg along the tibial nerve path. The TENS current parameters will be 200 microsecond pulse width, 10 Hz frequency, and intensity according to participant tolerance ranging between (10 - 50 mA) that increased gradually until visible movement in the big toe or fanning of toes will be noticed. The therapy sessions will be given three times a week, every other day, for a total of twelve sessions.
  Arms: study group (SG)
Device: Placebo Percutaneous Posterior Tibial Nerve Stimulation — placebo neuromodulation of the posterior tibial nerve in both lower limbs, much as those in the research group.
  Arms: control group (CG)
Behavioral: Home instructions — they will receive leaflet with information for home instructions on how to properly walk, sleep, maintain good posture, and deal with activities of daily living.

SUMMARY:
Background: Chronic pelvic pain (CPP) significantly impacts the quality of life in women. This study investigated the effects of transdermal neuromodulation in females with CPP.

Trial Design: Parallel, randomized, single-blind, controlled trial The aim of the study will be to examine the effect of posterior tibial nerve stimulation on women with idiopathic chronic pelvic pain syndrome.

Methods: Thirty females with chronic pelvic pain will be randomly allocated 1:1 to receive either transdermal neuromodulation of the posterior tibial nerve (intervention group) or advice to control posture (control group) for 4 weeks at the Outpatient Physical Therapy Clinic at Kafrelsheikh University in Egypt. The primary outcome was pain intensity measured by visual analog scale (VAS). Secondary outcomes were serum cortisol level and quality of life (QOL) score. Assessments will be done at baseline and after 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous, with a body mass index not exceeding 30 kg/m2 and complaining of idiopathic chronic pelvic pain syndrome (CPP).

Exclusion Criteria:

* chronic uterine prolapse, endometriosis, pelvic tumor, any sexual problems, an active genitourinary infection, heart diseases, kidney diseases, cognitive disorders or any physical or psychological condition that might impair the ability to provide written informed consent or adhere to the research procedure

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — indicate if participant eligibility is based on gender identity.
Enrollment: 35 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
VAS. | Before treatment and after 4 weeks of treatment
  measurement of pain level using visual analogue scale

SECONDARY OUTCOMES:
EQ-5D-5L | Before treatment and after 4 weeks of treatment
  EQ-5D-5L is a survey that will be used to evaluate health-related QOL
serum cortisol | Before treatment and after 4 weeks of treatment
  Early-morning serum cortisol concentration is an important biological marker for adequate pain control

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Kadry, PhD, Principal Investigator — Kafrelsheikh University
Locations (1):
- Kafrelshaikh University, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data from this study, including individual participant data (IPD) and associated documentation, will be made available upon reasonable request to the principal investigator. Requests will be considered when accompanied by a detailed proposal, including a clear justification for the use of the data. Such requests will be subject to a review process to ensure compatibility with participant consent and the ethical guidelines governing the study. Data sharing will be facilitated under a data use agreement that specifies the terms and conditions to ensure the privacy and confidentiality of participants
Supporting Information: Study Protocol, SAP
Time Frame: 1 year from publication
Access Criteria: Upon request from the principal investigator with appropriate justification